CLINICAL TRIAL: NCT03032068
Title: Feasibility of Home Monitoring After Primary Total Knee Arthroplasty
Brief Title: Home Monitoring After Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Staff Surgeon, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-1051
Record Dates: First submitted 2016-07-28; First posted 2017-01-26 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- At-Home Monitoring (Experimental): Patients will follow-up in clinic postoperatively at 4, 8, and 12 weeks and their recovery will also be monitored using sensors and communication devices while they are at home after surgery.
  Interventions: Other: At-Home Monitoring

INTERVENTIONS:
Other: At-Home Monitoring — Patient reported outcomes, functional measures such as the maximum attainable range of motion (AROM) and the number of steps taken will be tracked using sensors worn by the patient. The AROM sensor values will be verified with range of motion measurements taken using a goniometer during therapy and MD visits.

SUMMARY:
Home monitoring technologies have recently emerged in many different areas of healthcare. These technologies are being used to provide rehabilitation to patients, and to prevent, identify, and manage complications. The investigators are proposing a method to monitor and communicate with patients during the first 12 weeks after total knee arthroplasty (TKA) using an electronic home-based patient monitoring system with unique connectivity capabilities and prescriptive controls. The investigators will prospectively, electronically capture range of motion and gait parameters at specified intervals using Bluetooth sensors worn by the patient. The unique in-home patient monitoring platform will be utilized by 10 TKA patients once they return home following surgery. The investigators hypothesize that the use of an internet based home patient monitoring technology platform will reliably provide information related to the patients' pain and function and enhance patient feedback and communication after TKA. The hypothesis will be tested with the following aim: 1) To test the reliability of all technology utilized within the patient's home including but not limited to the sensors, the communication controller, the patient interface (Android tablet) and the internet by prospectively comparing between data collected through the home monitoring technology and traditional clinical measurements taken during physical therapy and surgical follow-up visits.

DETAILED DESCRIPTION:
Over one million primary total hip and total knee arthroplasty (TKA) surgeries are being performed annually in the U.S. and this number is expected to increase over the next seven years, along with a simultaneously projected shortage of trained orthopaedic surgeons to care for these patients. This proposal addresses the optimization of the surgeons' clinical time through utilization of innovative home based technologies to monitor and communicate with patients during the first 12 weeks after total knee arthroplasty. This will be accomplished by establishing home monitoring connectivity with novel technology and measure validated patient-reported outcomes, knee ROM and gait parameters in a postoperative TKA patient's native living environment. It will allow the investigators to prospectively, electronically capture clinically relevant TKA outcomes at the patient's home and provide insight into postoperative rehabilitation progress, predictors of suboptimal clinical outcomes, and guide future randomized controlled trial development to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary TKA
* Surgery is performed at Cleveland Clinic Main Campus or at Lutheran Hospital
* Patient must reside within 75 miles (driving distance) from Cleveland Clinic Main Campus
* Patient expected to utilize Cleveland Clinic Home Care Services after surgery

Exclusion Criteria:

* Revision or simultaneous bilateral TKA
* English is not the patient's preferred language for healthcare discussions
* Currently participating in any other research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Higuera, MD, Principal Investigator — Staff Surgeon
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were scheduled for primary total knee arthroplasty from October 2016 through February 2017 and met all enrollment criteria were asked to participate.
Pre-assignment Details: All participants were enrolled in the same group.
Groups:
- Home-based Monitoring: All enrolled patients were asked to use technology to collect functional and patient reported outcomes at home after total knee arthroplasty.
Period: Overall Study
Arm/Group | Home-based Monitoring
Started | 10
Preoperative Visit | 10
Postoperative Home Care Visit 1 | 10
Postoperative Home Care Visit 2 | 10
Postoperative Home Care Visit 3 | 10
4 Weeks Postoperative Visit | 9
8 Weeks Postoperative Visit | 9
12 Weeks Postoperative Visit | 9
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Patients who withdrew from the research prior to postoperative data collection were excluded from analysis. Therefore, these withdrawn patients do not have baseline information included here.
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 67 [61 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Reliability of Monitoring Technology, Measured as Proportion of Actual Data Received From the Patient's Home Compared to the Amount of Data Expected (Based on Activities That Were Reported as Completed by Patients) Over the 12 Week Study Period.
Description: The investigators will determine the reliability of the at-home monitoring technology for recording and transmitting data from the patient's home to the healthcare provider. This will be measured for each patient individually and then combined to form an aggregate measurement.
  Reliability of the technology to collect data was calculated for each patient individually by counting the number of times data (range of motion, TUG test results, VAS Pain score, etc) was received and dividing that number by the number of times data was expected (activities reported as complete by patients). This was then converted into a percentage. Additionally, this number was aggregated by combining the numerators (activities received) for all patients and denominators (activities complete) for all patients and determining the overall reliability of the technology.
Time Frame: daily, from the date of discharge until the 12 week postoperative follow-up appointment has occurred
Measure: Mean (Standard Deviation); unit: percentage of received vs expected data
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
percentage of received vs expected data | 91 (6)

2. Secondary Outcome: Rehab Compliance
Description: Percentage of required at-home therapy exercises completed each session, as well as the total percentage completed during all home therapy sessions
Time Frame: Percentage of exercises completed 2-3 times daily, from the date of discharge up to approximately 4 weeks postoperatively when outpatient physical therapy begins
Measure: Mean (Standard Deviation); unit: percentage of exercises completed
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
percentage of exercises completed
  Homecare Visit 2 | 88 (11)
  Homecare Visit 3 | 94 (7)
  4 Weeks Postop | 94 (13)

3. Secondary Outcome: Change From Preoperative to Postoperative Knee Range of Motion
Description: Change from Preoperative to Postoperative Knee Range of Motion, Knee range of motion is recorded daily using sensors above and below the knee. Please note: only data from sensors is being reported
Time Frame: Once preoperatively then postoperatively 2-3 times daily from the date of discharge until the 12 week postoperative follow-up appointment has occurred
Population: One patient was withdrawn from the study prior to the 8 week follow-up visit due to an adverse event. Therefore, only 9 patients were included in the analysis at 8 weeks and 12 weeks postoperative.
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
degrees
  Preoperative | 17 [4.2 to 29.8]
  Homecare Visit 1 | 5.8 [-18.5 to 30.2]
  Homecare Visit 2 | 9.7 [-8.6 to 28.0]
  Homecare Visit 3 | 2.2 [-42.3 to 46.7]
  4 Weeks Postoperative | -1.1 [-31.0 to 28.8]
  8 Weeks Postoperative: number analyzed (Participants) | 9
  8 Weeks Postoperative | 13.3 [-14.7 to 41.3]
  12 Weeks Postoperative: number analyzed (Participants) | 9
  12 Weeks Postoperative | 22.3 [11.3 to 33.3]

4. Secondary Outcome: Change From Preoperative to Postoperative Timed Up and Go Test
Description: Change from Preoperative to Postoperative Timed Up and Go Test. The time that a patient takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. This time was recorded electronically by the patient at home using the tablet.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: seconds difference
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
seconds difference
  Preoperative | 0.1 [-0.1 to 0.3]
  Homecare Visit 1 | 0.1 [-0.8 to 1.1]
  Homecare Visit 2 | 0.3 [-0.3 to 0.8]
  Homecare Visit 3 | 0.0 [-0.9 to 0.9]
  4 Weeks Postoperative | -0.3 [-1.2 to 0.7]
  8 Weeks Postoperative: number analyzed (Participants) | 9
  8 Weeks Postoperative | 0.6 [0.1 to 1.2]
  12 Weeks Postoperative | 0.2 [-0.1 to 0.6]

5. Secondary Outcome: Visual Analog Scale for Pain (Knee-related Pain at Its Worst Over a 24 Hour Period)
Description: Knee-related pain was measured using a visual analog scale with numeric values added to the line. Zero (0) is the minimum value and 10 is the maximum value. A score of 0 indicates no pain and a score of 10 indicates the worst pain imaginable.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
score on a scale
  Preoperative | 4 (3)
  Homecare Visit 1 | 4 (4)
  Homecare Visit 2 | 4 (2)
  Homecare Visit 3 | 4 (2)
  4 Weeks Postoperative | 4 (2)
  8 Weeks Postoperative: number analyzed (Participants) | 9
  8 Weeks Postoperative | 2 (2)
  12 Weeks Postoperative: number analyzed (Participants) | 9
  12 Weeks Postoperative | 1 (1)

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - KOOS Pain
Description: We will assess KOOS Pain using 9 questions, each response given a point value from 0 to 4. The sum of these points will total between 0 and 36 points. This score will be normalized to a 100 point scale where 100 means no pain and 0 is extreme pain.
Time Frame: Once preoperatively then postoperatively once weekly from the date of discharge until the 12 week follow-up appointment has occurred
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
score on a scale
  Preoperative | 41.7 (7.8)
  Homecare Visit 1 | 41.2 (10.0)
  Homecare Visit 2 | 54.6 (17.2)
  Homecare Visit 3 | 70.0 (5.0)
  4 Weeks Postoperative | 68.5 (16.3)
  8 Weeks Postoperative: number analyzed (Participants) | 9
  8 Weeks Postoperative | 73.7 (15.3)
  12 Weeks Postoperative: number analyzed (Participants) | 9
  12 Weeks Postoperative | 78.8 (11.6)

7. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - KOOS PS (Physical Function Short Form)
Description: We will assess KOOS Function using 7 questions, each response given a point value from 0 to 4. The sum of these points will total between 0 and 28 points. This total will be normalized to a 100 point scale where 100 means no functional difficulty and 0 is extreme difficulty.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
score on a scale
  Preoperative | 41.1 (12.7)
  Homecare Visit 1 | 36.3 (17.1)
  Homecare Visit 2 | 56.0 (18.0)
  Homecare Visit 3 | 62.8 (13.5)
  4 Weeks Postoperative | 73.0 (16.5)
  8 Weeks Postoperative: number analyzed (Participants) | 9
  8 Weeks Postoperative | 72.6 (16.2)
  12 Weeks Postoperative: number analyzed (Participants) | 9
  12 Weeks Postoperative | 78.1 (15.3)

8. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - KOOS QOL
Description: We will assess KOOS QOL using 4 questions, each response given a point value from 0 to 4. The sum of these points will total between 0 and 16 points, which will then be normalized to a 100 point scale. One hundred (100) means the knee does not affect quality of life and 0 indicates that the knee is a constant problem affecting quality of life.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Monitoring
Number analyzed (Participants) | 10
score on a scale
  Preoperative | 25.1 (8.8)
  Homecare Visit 1 | 25.0 (15.3)
  Homecare Visit 2 | 36.1 (12.8)
  Homecare Visit 3 | 43.8 (15.9)
  4 Weeks Postoperative | 50.0 (19.0)
  8 Weeks Postoperative: number analyzed (Participants) | 9
  8 Weeks Postoperative | 52.1 (14.0)
  12 Weeks Postoperative: number analyzed (Participants) | 9
  12 Weeks Postoperative | 57.8 (9.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through 12 weeks postoperatively for each participant.
Description: Adverse events were collected routinely at each follow-up visit during the study period
Arm/Group | Home-based Monitoring
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based Monitoring (N=14)
Quadriceps tendon tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Tore quadriceps tendon while getting into bed 2 weeks after surgery. This was not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT03032068/Prot_SAP_000.pdf